CLINICAL TRIAL: NCT02177240
Title: A Randomized Comparison of the Flex-it® Articulating Stylet to the GlideRite® Rigid Stylet for Orotracheal Intubation Using the GlideScope® in Simulated Difficult Intubations. A Double Blinded Randomized Controlled Trial.
Brief Title: A Comparison of the Flex-it® to the GlideRite® Stylet for GlideScope® in Simulated Difficult Intubations.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, John Viet Nguyen, MD, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Cér 14013
Record Dates: First submitted 2014-05-29; First posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Difficult Intubation
Keywords: GlideScope®; GlideRite®; Flex-it®; Difficult intubation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GRS (GlideRite®) (Active Comparator): GlideScope® intubation with GRS® stylet of a simulated difficult airway
  Interventions: Device: GlideScope® intubation with GRS® stylet
- FIS (Flex-it® ) (Active Comparator): GlideScope® intubation with Flex-it® stylet of a simulated difficult airway
  Interventions: Device: GlideScope® intubation with Flex-it® stylet

INTERVENTIONS:
Device: GlideScope® intubation with Flex-it® stylet — GlideScope® intubation with Flex-it® stylet of a simulated difficult airway
  Arms: FIS (Flex-it® )
Device: GlideScope® intubation with GRS® stylet — GlideScope® intubation with GRS® stylet of a simulated difficult airway
  Arms: GRS (GlideRite®)

SUMMARY:
The purpose of this study is to determine if the Flex-it® Articulating Stylet or the GlideRite® Rigid Stylet is more effective and less traumatic in the context of difficult GlideScope® intubations.

DETAILED DESCRIPTION:
Pre-operatively patient are approached and enrolled according to inclusion and exclusion criteria.

Demographic data is then recorded and afterwards the patient is randomized (randomization.com) but is blinded to the group.

The patient is outfitted with a Philadelphia® cervical collar and a BIS® monitor before induction of anesthesia.

The anesthetist is blinded to the randomization group. Once asleep, the patient is intubated using the GlideScope® with the single-use blade and one of the randomized intubation stylets by an operator.

Intubation and tube manipulation times, vital signs and BIS level are recorded via a nurse or video camera.

Verbal cues are given for start of laryngoscopy, tube manipulation and confirmation of CO2 which is recorded by the camera microphone.

Patient is questioned about hoarseness and sore throat when leaving the post anesthesia care unit according to our local protocol and 24hr after the surgical procedure.

The data is then taken from the video and analyzed by a blinded operator.

ELIGIBILITY:
Inclusion Criteria:

* ASA status 1-2
* BMI < 35
* Elective surgery
* General Anesthesia

Exclusion Criteria:

* Difficult intubation
* Indication for rapid sequence intubation
* Contraindication for cervical collar

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Intubation time | During intubation
  Time from start of laryngoscopy to confirmation of EtCO2

SECONDARY OUTCOMES:
Sore throat/Hoarseness | Day 0 (immediate post-operative)
  Scale of 0 to 3
Sore throat/Hoarseness | Day 1 (24hr post-operative)
  Scale of 0 to 3
Verbal Intubation difficulty scale | 15 minutes after intubation
  Scale of 1 to 10
Tube manipulation time | During Intubation
  Time from start of tube manipulation to confirmation of EtCO2
Resistance during stylet extraction | 15 minutes after intubation
  Scale of 1 to 5

CONTACTS AND LOCATIONS:
Overall Officials: John Viet Nguyen, MD, Principal Investigator — HMR; Issam Tanoubi, MD, Study Director — HMR
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada